CLINICAL TRIAL: NCT03258541
Title: TraceIT® Hydrogel Spacer Injections for Vagina and Erectile Bundles Sparing in Rectal Cancer Patients Treated With Neoadjuvant Radiotherapy: a Feasibility Study
Brief Title: Organ-sparing With TraceIT® for Rectal Cancer Radiotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Surgical access not facilitated- residues of hydrogel.
Sponsor: Thomas Zilli (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor-Investigator, Thomas Zilli, MD, PD, Médecin adjoint agrégé, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TraceIT_01268
Record Dates: First submitted 2017-05-17; First posted 2017-08-23 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Rectal Tumors; Rectal Cancer; Advanced Cancer
Keywords: TraceIT®; Hydrogel spacer; Rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: TraceIT® — This pilot study wishes to investigate feasibility and efficacy of the injected hydrogel spacers TraceIT® in sparing vagina/prostate in the treatment of rectal cancer patients.
Radiation: Volumetric Arc Therapy (VMAT) — VMAT - fractionation Schedule : 1.8 Gy per fraction, one fraction per day, 5 fractions per week for the elective PTV and 2 Gy per fraction, one fraction per day, 5 fractions per week for the PTV-boost using a simultaneous integrated boost technique.
Procedure: Surgery — Low anterior resection of the rectum: 8-10 weeks post-radiotherapy

SUMMARY:
For advanced rectal tumors, the standard of care is neoadjuvant radiotherapy (RT) +/- chemotherapy followed by surgery 8-10 weeks later. Despite its proven efficacy in reducing local relapse, the neo-adjuvant treatment has been associated to non-negligible side effects, especially in terms of impaired sexual function. For females, pelvic RT is frequently associated to long-term complications such as vaginal stenosis (VS), vaginal dryness, and dyspareunia, while in men RT doses delivered to the neurovascular peri-prostatic bundles and penile bulb have been associated to the risk to develop erectile dysfunction.

In prostate cancer, hydrogel spacers have been evaluated to create space between the target (prostate) and the organ (rectum) to be spared during radiotherapy treatments. Clinical studies have shown the ease of spacer application; patient tolerance and, good clinical outcomes (decrease in rectal toxicities).

This pilot study wishes to investigate feasibility and efficacy of the injected hydrogel spacers TraceIT® in sparing vagina/prostate in the treatment of rectal cancer patients.

DETAILED DESCRIPTION:
This is a feasibility prospective pilot study. Ten patients (5 males and 5 females) with a histologically proven locally advanced rectal cancer with the indication of neoadjuvant radiotherapy or radio-chemotherapy will be recruited for this study. Prior to enrollment, potential candidates will undergo a thorough physical and clinical examination and documentation on medical and surgical history. If eligible, a baseline planning computed tomography (CT) simulation will be performed at the Radiation Oncology Department before the TraceIT® implant. Participants will undergo a transperineal injection of TraceIT® spacer gel between rectum and vagina or prostate performed by a trained radiologist under transrectal ultrasound guidance. A CT simulation will be repeated within 3 to 5 days post injection using the same imaging modality and treatment position used the pre- TraceIT® injection. Radiation treatment plans will be generated using scans realized pre- and post- TraceIT® injection and compared using dose volume histograms (DVH) analyses. Tolerance, side effects, and adverse events related to the procedure will be recorded prospectively from the injection until week-4 after EBRT (External Beam Radiation Therapy) completion. Radiological status of the spacer will be evaluated on the preoperative magnetic resonance Imaging (MRI). Histopathological results and any serious and/or unanticipated adverse events following surgery procedure will be recorded retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* WHO (World Health Organization) performance status 0-1 at registration
* Locally advanced (T1-2 node positive or T3 N0/N+) histologically proven rectal adenocarcinoma located in the middle or in the high rectum. Patients with tumors located in the lower rectum may be eligible if the location of the tumor do not preclude the implant of the spacer (i.e. tumors located anteriorly in the proximity of the anal sphincter)
* Indication for preoperative radiotherapy or radio-chemotherapy
* Absence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration/randomization, written informed consent must be given according to GCP/ICH (Guideline for Good Clinical Practice/Harmonised Tripartite Guideline), and national/local regulations.

Exclusion Criteria:

* Patient <18 years old
* WHO performance status ≥ 2 at registration
* Patient with a local extension, clinical stage T4 and/or presenting a vagina/prostate/bladder invasion
* Active bleeding disorder or clinically significant coagulopathy (PTT >35sec/ or INR >1.4 (INR, international normalized ratio). Or platelet count < 100'000/mm3)
* Active inflammatory or infectious process involving the perineum, gastrointestinal or urinary tract
* Compromised immune system (e.g. HIV/acquired immunodeficiency syndrome, autoimmune disease or immunosuppressive therapy)
* History of previous pelvic surgery
* History of active inflammatory bowel disease (Crohn's disease, ulcerative colitis, irritable bowel disease)
* Contraindication for MRI
* Pregnant or lactating females
* Inability to provide a written informed consent
* Inability to comply with study and follow up procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Clinical performance | 2 years
  Incidence of serious adverse events.

SECONDARY OUTCOMES:
Comparative dosimetric studies | 2 years
  Dosimetric parameters to determine effectiveness of this technique to reduce RT (radiotherapy) doses to the vagina/erectile bundles as assessed by comparative dosimetric studies.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No